CLINICAL TRIAL: NCT00640809
Title: Double-Blind, Placebo-Controlled, Randomized Two-Week Study, Comparing Small Bowel Lesions Associated With Celecoxib (200 mg BID) vs. Ibuprofen (800 mg TID) Plus Omeprazole (20 mg QD)
Brief Title: Comparison of Small Bowel Lesions Associated With Celecoxib Versus Ibuprofen Plus Omeprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191071
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Bowel Diseases, Inflammatory
Keywords: Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Intestinal Diseases | interventions — Celecoxib; Ibuprofen; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Placebo Comparator)
  Interventions: Other: Placebo
- C (Active Comparator)
  Interventions: Drug: Ibuprofen plus Omeprazole

INTERVENTIONS:
Drug: Celecoxib — 200 mg oral capsule twice daily for 2 weeks
  Arms: A
Other: Placebo — Matched placebo for 2 weeks
  Arms: B
Drug: Ibuprofen plus Omeprazole — ibuprofen 800 mg oral tablet three times daily plus omeprazole 20 mg oral capsule once daily for 2 weeks
  Arms: C

SUMMARY:
To evaluate the small bowel lesion pattern associated with celecoxib alone versus ibuprofen plus omeprazole

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Normal, healthy gastrointestinal tract (no small bowel mucosal breaks at Day 14 according to endoscopic data
* No history of GI ulcers, bleeding or surgery, or complete or partial stenosis of the small intestine
* Willing not to drink any alcohol during study period

Exclusion Criteria:

Exclusion criteria:

* Has established delayed gastric emptying or diabetic gastroparesis
* Has active gastroesophageal reflux disease or requires anti-ulcer medications
* Has taken aspirin or nonsteroidal antinflammatory drugs (ibuprofen, naproxen) more than 3 times per week within 2 weeks prior to the screening visit; aspirin for cardiovascular prophylaxis is restricted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2003-10; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Number of mucosal breaks in the small bowel for each subject | Day 30

SECONDARY OUTCOMES:
Adverse events | Day 30
Laboratory tests | Day 30
Vital signs | Day 30
Correlation of number of mucosal breaks in the small bowel for each patient with the result of the fecal calprotectin test | Day 30
Percentage of subjects with gastric mucosal breaks and the number of mucosal breaks | Day 30
Change from screening visit in hemoglobin and hematocrit | Day 30
Correlation of the number of gastric mucosal breaks with the number of small bowel mucosal breaks | Day 30
Physical examination | Day 30
Percentage of subjects with >=1 mucosal breaks | Day 30
Total number of small bowel lesions with or without hemorrhage | Day 30
Percentage of subjects with visible blood in the small bowel (without visualized lesions in the small bowel) | Day 30
Change in Patient General Questionnaire Visual Analog Scale from Day 16 | Day 30
Change in Severity of Dyspepsia Assessment questionnaire from Day 16 | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191071&StudyName=Comparison%20of%20Small%20Bowel%20Lesions%20Associated%20with%20Celecoxib%20versus%20Ibuprofen%20Plus%20Omeprazole